CLINICAL TRIAL: NCT03793972
Title: Triaging and Referring in Adjacent General and Emergency Departments (the TRIAGE-trial): a Cluster Randomised Controlled Trial
Brief Title: Triaging and Referring in Adjacent General and Emergency Departments
Acronym: TRIAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Veronique Verhoeven, Principal Investigator, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: T000718N
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Triage
Keywords: Triage; Primary Health Care; Emergency Service, Hospital
MeSH Terms: conditions — Emergencies | interventions — Triage

STUDY DESIGN:
Intervention Model Description: Cluster randomised with weekends servings as clusters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triage with referral to primary care (Experimental): Triage and referral according to eMTS.
  Interventions: Other: Triage with referral to primary care
- Triage without referral to primary care (Active Comparator): Weekends with usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Triage with referral to primary care — During intervention weekends(and holidays) a nurse will triage patients using a newly developped extended Manchester Triage System (eMTS). Patients appropriate for primary care will be referred to the general practitioner on call.We will inform patients about the nature of the intervention using leaflets and broadcasting in the waiting room of the Emergency Department.
  Arms: Triage with referral to primary care
Other: Usual care — During a control weekend (and holidays), all data registration and collection will be the same as during intervention weekends but patents will not be informed about their allocation advice. The emergency physician will see all patients deciding to stay at the ED, without influence of the triage advice. As in standard clinical care, patients will have the right to change their mind and go spontaneously to the general practitioner. . During control weekends, we will only inform about triage in general but no about the general practioner or the intervention.
  Arms: Triage without referral to primary care

SUMMARY:
Introduction: Patients who might also go to the general practitioner (GP) frequently consult emergency departments (ED). This leads to additional costs for both government and patient and a high workload for emergency physicians in Flanders. The Belgian government wants to address this problem by improved collaboration between EDs and general practice cooperatives (GPCs).

Intervention: Patients presenting at the ED during out-of-hours (OOH) will be triaged and allocated to the most appropriate service. For this purpose the Manchester Triage System (MTS) which is commonly used in Flemish hospitals, will be extended (eMTS). By doing so a trained nurse will be able to diverge suitable patients towards the GPC.

Methodology: The investigators will conduct a cluster randomised controlled trial in which eligible ED patients will be diverged to the GPC using the eMTS. The investigators will collect data using the iCAREdata database. The investigators will study the use of the eMTS, the effectiveness and effects of triage, work load changes, epidemiology at both departments, patient safety, health insurance (HIS) and patient expenditures. Furthermore, facilitators and barriers will be studied and an incident analysis of problem cases will be performed.

Outcome: The primary outcome is the proportion of patients who enter the ED and are handled by the GP after triage. Secondary outcome measurements are related to safety: referral rate to the ED by the GP, proportion of patients not following the triage advice and file review for selected patients.

ELIGIBILITY:
Inclusion Criteria:

* availability of a Belgian citizen national insurance number

Exclusion Criteria:

* Patients arriving at the ED by an ambulance with a doctor or nurse
* Patients all ready admitted to an other hospital department

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8158 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Verhoeven, PhD, Principal Investigator — Univeristeit Antwerpen
Locations (2):
- Belgium (2):
  - AZ Monica, Deurne
  - HuisartsenWachtpost Antwerpen Oost, Deurne

IPD SHARING:
Plan to Share IPD: No
Even the researchers will only have very limited access to individual data. All collected data will be stored in the "iCAREdata" database (see http://www.icaredata.eu/) and as such will be accessible when necessary.

REFERENCES:
- [Derived] Morreel S, Verhoeven V, Philips H, Meysman J, Homburg I, De Graeve D, Monsieurs KG. Differences in emergency nurse triage between a simulated setting and the real world, post hoc analysis of a cluster randomised trial. BMJ Open. 2022 Jul 1;12(7):e059173. doi: 10.1136/bmjopen-2021-059173. PMID 35777880
- [Derived] Homburg I, Morreel S, Verhoeven V, Monsieurs KG, Meysman J, Philips H, De Graeve D. Non-compliance with a nurse's advice to visit the primary care provider: an exploratory secondary analysis of the TRIAGE-trial. BMC Health Serv Res. 2022 Apr 8;22(1):463. doi: 10.1186/s12913-022-07904-8. PMID 35395840
- [Derived] Morreel S, Philips H, De Graeve D, Monsieurs KG, Kampen JK, Meysman J, Lefevre E, Verhoeven V. Triaging and referring in adjacent general and emergency departments (the TRIAGE trial): A cluster randomised controlled trial. PLoS One. 2021 Nov 3;16(11):e0258561. doi: 10.1371/journal.pone.0258561. eCollection 2021. PMID 34731198

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Weekends
Period: Overall Study
Arm/Group | Triage With Referral to Primary Care | Triage Without Referral to Primary Care
Started | 6374; 37 Weekends | 1784; 10 Weekends
Completed | 6374; 37 Weekends | 1784; 10 Weekends
Not Completed | 0; 0 Weekends | 0; 0 Weekends

BASELINE CHARACTERISTICS:
Population: See main publication for details.
Groups:
- Total: Total of all reporting groups
Arm/Group | Triage With Referral to Primary Care | Triage Without Referral to Primary Care | Total
Number analyzed (Participants) | 6374 | 1784 | 8158
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (25) | 39 (24) | 38 (25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3149 | 880 | 4029
  Male | 3225 | 904 | 4129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6374 | 1784 | 8158

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Presenting at the ED But Being Treated by the GPC After Referral
Description: The difference between intervention and control period will be calculated. Treatment at the GPC means having a record at the GPC.
Time Frame: Patient flow will be followed for 24 hours after presentation at the ED
Population: See main paper for more details.
Measure: Count of Participants; unit: Participants
Arm/Group | Triage With Referral to Primary Care | Triage Without Referral to Primary Care
Number analyzed (Participants) | 6294 | 1744
Participants | 599 | 0

ADVERSE EVENTS:
Time Frame: For the individual patient: only during their stay at the emergency department or general practice cooperative.
Description: Due to the nature of the intervention, no systematic system for adverse events was used. See main paper for what was used in practice.
Arm/Group | Triage With Referral to Primary Care | Triage Without Referral to Primary Care
All-Cause Mortality (participants affected / at risk) | 1/6294 | 0/1744
Serious Adverse Events (participants affected / at risk) | 1/6294 | 0/1744
Other Adverse Events (participants affected / at risk) | 0/6294 | 0/1744
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triage With Referral to Primary Care (N=6294) | Triage Without Referral to Primary Care (N=1744)
Ruptured Abdominal Aortic Artery (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — see main paper

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT03793972/Prot_SAP_000.pdf